CLINICAL TRIAL: NCT02336165
Title: Phase 2 Study to Evaluate the Clinical Efficacy and Safety of MEDI4736 in Patients With Glioblastoma (GBM)
Brief Title: Phase 2 Study of Durvalumab (MEDI4736) in Patients With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: MedImmune LLC (Industry); Cancer Research Institute, New York City (Other); Cure Brain Cancer Foundation, Australia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2013-006
Record Dates: First submitted 2014-12-23; First posted 2015-01-12 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Immunotherapy; T Cell; PD-L1; MEDI4736; Radiation; Radiotherapy; GBM
MeSH Terms: conditions — Glioblastoma | interventions — durvalumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A (Experimental): Subjects with newly diagnosed unmethylated MGMT GBM receive durvalumab (10 mg/kg Q2W) + standard radiotherapy.
  Interventions: Drug: Durvalumab; Radiation: Standard radiotherapy
- Cohort B (Experimental): Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) as monotherapy.
  Interventions: Drug: Durvalumab
- Cohort B2 (Experimental): Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) + bevacizumab (10 mg/kg Q2W).
  Interventions: Drug: Durvalumab; Biological: Bevacizumab
- Cohort B3 (Experimental): Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) + bevacizumab (3 mg/kg Q2W).
  Interventions: Drug: Durvalumab; Biological: Bevacizumab
- Cohort C (Experimental): Bevacizumab-refractory subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) + continued bevacizumab (10 mg/kg Q2W).
  Interventions: Drug: Durvalumab; Biological: Bevacizumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is administered as an IV infusion over 60 ± 5 minutes Q2W.
  Other Names: MEDI4736
Radiation: Standard radiotherapy — Focal radiotherapy is administered at 2 Gy given daily 5 days per week for a total of 60 Gy over 30 fractions per local institutional guidelines or local prescribing information. On days when radiotherapy and durvalumab overlap, radiotherapy is administered first followed by durvalumab.
  Arms: Cohort A
Biological: Bevacizumab — Bevacizumab is administered as an IV infusion (per local prescribing information) Q2W. When durvalumab and bevacizumab are administered together (i.e., Cohorts B2, B3, and C), durvalumab is administered first followed by a 1-hour observation period, after which, bevacizumab is infused.
  Other Names: Avastin
  Arms: Cohort B2; Cohort B3; Cohort C

SUMMARY:
This is an ongoing Phase 2, open-label, multicenter, non-randomized study of MEDI4736 (durvalumab) in subjects with glioblastoma (GBM) enrolled into 5 non-comparative cohorts. Primary study objectives, which vary by cohort due to differences in subject populations, include evaluation of the clinical efficacy as measured by the overall survival (OS) rate at 12 months (Cohort A), progression-free survival (PFS) at 6 months (Cohorts B, B2, and B3), and OS at 6 months (Cohort C). For all cohorts, secondary objectives include evaluation of the safety/tolerability and clinical efficacy of study treatment, and exploratory objectives include evaluation of the neurologic function and correlative biomarkers.

DETAILED DESCRIPTION:
Eligible subjects are enrolled in parallel into one of the following 5 cohorts as described below. In each cohort, the first study drug administration for the first subject and the second subject are separated by at least 1 week.

* Cohort A: Subjects with newly diagnosed unmethylated O^6-methylguanine-deoxyribonucleic acid methyltransferase (MGMT) GBM receive durvalumab (10 mg/kg every 2 weeks [Q2W]) + standard radiotherapy. The first 6 subjects are evaluated for dose-limiting toxicity (DLT) for 10 weeks to determine whether the durvalumab dose should be lowered to 3 or 1 mg/kg.
* Cohort B: Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) as monotherapy.
* Cohort B2: Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) + bevacizumab (10 mg/kg Q2W).
* Cohort B3: Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) + bevacizumab (3 mg/kg Q2W).
* Cohort C: Bevacizumab-refractory subjects with recurrent GBM receive durvalumab (10 mg/kg Q2W) + continued bevacizumab (10 mg/kg Q2W). The first 6 subjects are evaluated for DLTs for 6 weeks to determine whether the durvalumab dose should be lowered to 3 or 1 mg/kg.

The Core Study lasts for up to 12 months; optional extension treatment may be offered to subjects who complete 51 weeks of treatment on the Core Study with stable disease or better and upon agreement between the subject, Investigator, and Sponsor.

Subjects are followed on study for 90 days after the last drug administration and off study every 6 months for 3 years from the date of the first dose of study treatment.

The primary study endpoints have been met, although some subjects remain in treatment and/or follow-up and data collection is ongoing.

ELIGIBILITY:
Inclusion Criteria [criteria apply to all cohorts unless otherwise specified]:

1. Cohort A: Subjects with newly diagnosed, untreated, unmethylated MGMT GBM who are eligible for standard radiation therapy.
2. Cohorts B, B2, B3 and C: First or second recurrence of GBM by diagnostic biopsy or contrast enhanced magnetic resonance imaging (MRI) per modified Response Assessment in Neuro-oncology (RANO) criteria, with last baseline MRI confirmation within 14 days prior to Study Day 1. Note: Recurrence is defined as progression following therapy (i.e., chemotherapy; radiation). If the subject had a surgical resection for relapsed disease and no anti-tumor therapy was administered for up to 12 weeks, and the subject has further evidence of tumor growth or undergoes another resection, this will be considered as one episode of recurrence.
3. Cohorts B, B2, B3 and C: On Study Day 1, at least 12 weeks from prior radiotherapy (unless progressive disease outside of the radiation field or histopathologic confirmation of unequivocal tumor).
4. Cohorts B, B2, B3: No prior vascular endothelial growth factor (VEGF)/VEGF receptor targeted therapy; Cohort C: No more than one prior bevacizumab regimen.
5. Cohorts B, B2, B3 and C: Recovery from any prior treatment clinically significant, related adverse events to grade ≤ 1 or pretreatment baseline with the exception of alopecia and laboratory values listed per inclusion criteria.
6. Subjects with measurable or non-measurable disease.
7. Histopathologic confirmation of glioblastoma.
8. At the time of Study Day 1, subjects must be at least 4 weeks since major surgical procedure, open biopsy, or significant traumatic injury; there should be no anticipation of need for major surgical procedure during the course of the study. There should be no core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Study Day 1.
9. Subjects who have previously been treated with the Optune™ device are eligible for the study as long as toxicity related to the treatment has resolved to ≤ grade 1 or baseline.
10. Eastern Cooperative Oncology Group (ECOG) ≤ 1 or Karnofsky performance status of ≥ 70.
11. Adequate hematologic, renal and hepatic function, as defined below:

    * Absolute neutrophil count ≥ 1000/mm^3;
    * Platelet count ≥ 100,000/mm^3;
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN); or if subject has Gilbert syndrome, then total bilirubin ≤ 3 x ULN;
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 x ULN;
    * Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 50 mL/min (using the Cockcroft-Gault formula):

      * Female CrCl = (140 - age in years) x weight in kg x 0.85/72 x serum creatinine in mg/dL;
      * Male CrCl = (140 - age in years) x weight in kg x 1.00/72 x serum creatinine in mg/dL;
    * Cohorts B2, B3 and C: Urinary protein quantitative value of ≤ 30 mg/dL in urinalysis or ≤1+ on dipstick, unless quantitative protein is < 1000 mg in a 24-hour urine sample.
12. Age must be greater than or equal to 18 years at date of consent.
13. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria [criteria apply to all cohorts unless otherwise specified]:

1. Primary tumors localized to the brain stem or spinal cord.
2. Locally directed therapies including but not limited to stereotactic radiosurgery, re-irradiation, Gliadel®, and therapeutics administered by direct injection or convection-enhanced delivery within 6 months of start of study treatment.
3. Prior exposure to durvalumab or other programmed cell death-1 (PD-1), programmed cell death ligand-1 (PD-L1), cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibodies.
4. Presence of diffuse leptomeningeal disease or extracranial disease.
5. Active, suspected or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, irritable bowel syndrome, Wegner's granulomatosis and Hashimoto's thyroiditis). Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
6. Known primary immunodeficiency or active human immunodeficiency virus.
7. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months indicated by positive test for hepatitis B virus surface antigen or hepatitis C virus ribonucleic acid (hepatitis C virus antibody).
8. History of organ transplant requiring use of immunosuppressive medication.
9. History of active tuberculosis.
10. Significant active systemic illness including infections requiring intravenous antibiotics.
11. Current pneumonitis or interstitial lung disease.
12. Other invasive malignancy within 2 years prior to entry into the study, except for those treated with surgical therapy only.
13. History of severe allergic reactions to any unknown allergens or any components of the study drugs.
14. Any prior grade ≥ 3 immune-related adverse event (irAE) or any prior corticosteroid-refractory irAE.
15. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
16. Lack of availability for follow-up assessments.
17. Lack of availability for Post Study Follow-up contacts to determine relapse and survival.
18. Women who are breast-feeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin).
19. Women of childbearing potential not using a medically acceptable means of contraception for the duration of the study and unsterilized males not willing to abide by protocol-specified requirements for contraception.
20. If a subject previously received another investigational treatment, the last dose of investigational treatment was administered within 4 weeks of Day 1 of the study.
21. Any condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.
22. Cohorts B2, B3, and C:

    * Evidence of hemorrhage on the baseline MRI or computed tomography (CT) scan other than those that are ≤ grade 1 and either post-operative or stable on at least two consecutive scans;
    * Current use of warfarin sodium or any other Coumadin®-derivative anticoagulant. Participant must be off Coumadin-derivative anticoagulants for at least 7 days prior to starting study drug. Low molecular weight heparin and Factor Xa antagonists are allowed;
    * History of clinically significant bleeding within 6 months of enrollment;
    * History of arterial thromboembolism within 12 months prior to enrollment;
    * Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications);
    * Any prior history of hypertensive crisis or hypertensive encephalopathy;
    * Clinically significant cardiovascular disease within 12 months prior to enrollment (or randomization), including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent;
    * Evidence of bleeding diathesis or coagulopathy;
    * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment;
    * Serious, non-healing wound, ulcer, or bone fracture.
23. Subjects must not donate blood while on study and for at least 90 days following the last durvalumab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Study Chair — Dana-Farber Cancer Institute
Locations (7):
- United States (6):
  - Research Facility, Los Angeles, California
  - Research Facility, San Francisco, California
  - Research Facility, Baltimore, Maryland
  - Research Facility, Boston, Massachusetts
  - Research Facility, St Louis, Missouri
  - Research Facility, New York, New York
- Research Facility, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giesinger JM, Kieffer JM, Fayers PM, Groenvold M, Petersen MA, Scott NW, Sprangers MA, Velikova G, Aaronson NK; EORTC Quality of Life Group. Replication and validation of higher order models demonstrated that a summary score for the EORTC QLQ-C30 is robust. J Clin Epidemiol. 2016 Jan;69:79-88. doi: 10.1016/j.jclinepi.2015.08.007. Epub 2015 Sep 28. PMID 26327487

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Subjects with newly diagnosed unmethlyated O^6-methylguanine-deoxyribonucleic acid methyltransferase (MGMT) glioblastoma (GBM) receive durvalumab (10 mg/kg IV Q2W) + standard radiotherapy (2 Gy/day x 5 days per week, for a total of 60 Gy over 30 fractions per local guidelines). On days when radiotherapy and durvalumab overlap, radiotherapy is administered first followed by durvalumab.
- Cohort B: Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg IV Q2W) as monotherapy.
- Cohort B2: Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg IV Q2W) + bevacizumab (10 mg/kg IV Q2W).
  Durvalumab is administered first followed by a 1-hour observation period, after which, bevacizumab is infused.
- Cohort B3: Bevacizumab-naïve subjects with recurrent GBM receive durvalumab (10 mg/kg IV Q2W) + bevacizumab (3 mg/kg IV Q2W).
  Durvalumab is administered first followed by a 1-hour observation period, after which, bevacizumab is infused.
- Cohort C: Bevacizumab-refractory subjects with recurrent GBM receive durvalumab (10 mg/kg IV Q2W) + continued bevacizumab (10 mg/kg IV Q2W).
  Durvalumab is administered first followed by a 1-hour observation period, after which, bevacizumab is infused.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Started | 40 | 31 | 33 | 33 | 22
Completed | 6 | 6 | 2 | 2 | 0
Not Completed | 34 | 25 | 31 | 31 | 22
Not completed — Death | 3 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 2 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 4 | 1 | 2 | 4 | 1
Not completed — Progressive disease | 23 | 22 | 27 | 24 | 19
Not completed — Non-compliance | 1 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population comprises all subjects who received any dose of durvalumab.
Groups:
- Cohort A: Subjects with newly diagnosed unmethlyated MGMT GBM receive durvalumab (10 mg/kg IV Q2W) + standard radiotherapy (2 Gy/day x 5 days per week, for a total of 60 Gy over 30 fractions per local guidelines). On days when radiotherapy and durvalumab overlap, radiotherapy is administered first followed by durvalumab.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C | Total
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22 | 159
Age, Continuous [Median (Full Range); unit: years] | 57.0 [22 to 77] | 54.0 [24 to 77] | 57.0 [40 to 74] | 54.0 [23 to 73] | 56.5 [37 to 77] | 56.0 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 15 | 13 | 8 | 53
  Male | 28 | 26 | 18 | 20 | 14 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 38 | 27 | 28 | 30 | 19 | 142
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 4 | 2 | 1 | 13
Region of Enrollment [Number; unit: participants]
  United States | 38 | 30 | 33 | 33 | 21 | 155
  Australia | 2 | 1 | 0 | 0 | 1 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    ECOG PS 0 | 24 | 16 | 9 | 10 | 6 | 65
    ECOG PS 1 | 16 | 15 | 24 | 23 | 16 | 94
O^6-Methylguanine Deoxyribonucleic Acid Methyltransferase (MGMT) Methylation Status [Count of Participants; unit: Participants]
  Methylated | 0 | 9 | 12 | 12 | 9 | 42
  Unmethylated | 40 | 15 | 18 | 18 | 11 | 102
  Unknown | 0 | 7 | 3 | 3 | 2 | 15
Isocitrate dehydrogenase (IDH) Mutation Status [Count of Participants; unit: Participants]
  IDH Mutant | 5 | 4 | 4 | 2 | 1 | 16
  Wild Type | 35 | 22 | 28 | 30 | 19 | 134
  Unknown | 0 | 5 | 1 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 12 Months (OS-12) as Estimated Using the Kaplan-Meier Method (Cohort A)
Description: OS-12 with 90% confidence interval (CI) is the primary endpoint of Cohort A and is the percentage of subjects who remain alive at 12 months, where OS is measured from the time of diagnosis until the recorded date of death or last follow-up. Subjects who are lost to follow-up at the time of the analysis will be censored on the date of last follow-up.
Time Frame: Up to 12 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Number (90% Confidence Interval); unit: percent of subjects alive
Arm/Group | Cohort A
Number analyzed (Participants) | 40
percent of subjects alive | 60.0 [46.1 to 71.4]

2. Primary Outcome: Progression-free Survival Rate at 6 Months (PFS-6) as Estimated Using the Kaplan-Meier Method (Cohorts B, B2, and B3)
Description: PFS-6 is the primary endpoint of Cohorts B, B2, and B3, and is the percentage of subjects who have not progressed at 6 months, with PFS measured from the date of the first dose of study treatment to the date of earliest disease progression (PD) based on modified Response Assessment in Neuro-Oncology (RANO) criteria or to the date of death, if PD does not occur. Per the RANO criteria, PD indicates any new lesion or a 25% increase in sum of the products of perpendicular diameters of enhancing lesions, or clear clinical deterioration per the Investigator (Wen et al. J Clin Oncol 2010; 28(11):1963-72).
Time Frame: Up to 6 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B | Cohort B2 | Cohort B3
Number analyzed (Participants) | 31 | 33 | 33
percentage of participants | 19.4 [9.3 to 32.1] | 15.2 [6.7 to 26.8] | 17.2 [7.7 to 29.7]

3. Primary Outcome: Overall Survival Rate at 6 Months (OS-6) as Estimated Using the Kaplan-Meier Method (Cohort C)
Description: OS-6 is the primary endpoint of Cohort C and is the percentage of subjects who remain alive at 6 months, where OS is measured from the date of the first dose of study treatment until the recorded date of death or last follow-up. Subjects who are lost to follow-up at the time of the analysis will be censored on the date of last follow-up.
Time Frame: Up to 6 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C
Number analyzed (Participants) | 22
percentage of participants | 36.4 [23.5 to 49.3]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) are reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, magnetic resonance imaging, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 90 days after the last dose of durvalumab. AEs are considered to be treatment emergent if they occur or worsen in severity after the first dose of study treatment.
Time Frame: Up to 15 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22
Participants
  Any TEAE | 40 | 31 | 33 | 33 | 22
  Serious TEAE | 26 | 18 | 11 | 15 | 14
  Treatment-related TEAE | 37 | 26 | 30 | 31 | 17

5. Secondary Outcome: Median PFS as Estimated Using the Kaplan-Meier Method
Description: PFS is measured from the date of the first dose of study treatment to the date of earliest PD based on modified RANO criteria or to the date of death, if PD does not occur. Per the RANO criteria, PD indicates any new lesion or a 25% increase in sum of the products of perpendicular diameters of enhancing lesions, or clear clinical deterioration per the Investigator (Wen et al. J Clin Oncol 2010; 28(11):1963-72).
Time Frame: Up to 15 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22
weeks | 19.9 [16.0 to 32.3] | 13.0 [7.4 to 20.1] | 16.0 [11.9 to 16.1] | 15.7 [8.3 to 16.4] | 7.9 [5.3 to 8.6]

6. Secondary Outcome: Median OS as Estimated Using the Kaplan-Meier Method
Description: All subjects are followed for survival at least every 6 months for up to 3 years following initiation of study treatment. In Cohort A, OS is measured from the date of diagnosis until the recorded date of death or last follow-up. In Cohorts B, B2, B3, and C, OS is measured from the date of the first dose of study treatment until the recorded date of death or last follow-up. Subjects who remain alive or are lost to follow-up at the time of the analysis are censored on the date of last follow-up.
Time Frame: Up to 36 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22
weeks | 64.8 [51.6 to 78.9] | 39.4 [23.7 to 64.3] | 37.3 [24.4 to 43.4] | 39.7 [26.9 to 47.4] | 19.3 [10.3 to 27.7]

7. Secondary Outcome: Number of Subjects With Best Overall Response
Description: Radiographic response is assessed by consistent imaging methods every (q) 8 to 9 weeks during study treatment administration. Response is categorized per the modified RANO criteria: complete response (CR) indicates no new lesions and disappearance of all disease sustained for ≥ 4 weeks; partial response (PR) indicates no new lesions, no progression of non-measureable disease, and ≥ 50% decrease from baseline in sum of products of perpendicular diameters of measurable lesions sustained for ≥ 4 weeks; stable disease (SD) indicates non-qualification for CR, PR, or progressive disease (PD); PD indicates any new lesion or a 25% increase in sum of the products of perpendicular diameters of enhancing lesions, or clear clinical deterioration per the Investigator (Wen et al. J Clin Oncol 2010; 28(11):1963-72).
Time Frame: Up to 15 months
Population: The population comprises all subjects who received any dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22
Participants
  CR | 1 | 0 | 0 | 0 | 0
  PR | 4 | 4 | 3 | 3 | 0
  SD | 26 | 12 | 20 | 18 | 6
  PD | 9 | 15 | 10 | 11 | 14
  Unknown Response | 0 | 0 | 0 | 1 | 2

8. Secondary Outcome: Mean Changes From Baseline in the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30)
Description: Health-related quality of life was measured using the validated EORTC-QLQ-C30. Questionnaires may be completed by the subject or with the assistance of the examiner at baseline prior to initiation of study therapy, and then approximately every 8 weeks while on study treatment (prior to discussing treatment response at each visit, whenever possible).
  All questions are answered using a categorical scale (1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much for symptoms and 1= very poor; 7= excellent for global heath questions). Scores were linearly transformed to 0 to 100 scales so that higher scores represented a higher level of functioning.
  Overall scores were calculated for each patient for each timepoint (Giesinger J et al Journal of Clinical Epidemiology. 2016 Jan;69:79-88). Mean change from baseline where baseline is the last non-missing value before the administration of MEDI4736 was reported.
Time Frame: Up to 12 months
Population: Number of subjects who completed European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) at baseline and each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22
units on a scale
  Week 9: number analyzed (Participants) | 29 | 15 | 24 | 26 | 10
  Week 9 | -6.03 (19.53) | -8.33 (26.16) | -5.56 (21.80) | -7.05 (20.78) | -12.50 (24.30)
  Week 17: number analyzed (Participants) | 25 | 8 | 14 | 14 | 4
  Week 17 | -2.0 (18.05) | 4.17 (27.46) | -7.14 (26.53) | -7.74 (18.62) | -16.67 (6.80)
  Week 25: number analyzed (Participants) | 20 | 4 | 9 | 5 | 0
  Week 25 | 0.42 (15.64) | 10.42 (17.18) | -3.70 (31.49) | -8.33 (19.54) |
  Week 33: number analyzed (Participants) | 8 | 3 | 4 | 3 | 0
  Week 33 | -6.25 (15.27) | 30.56 (20.97) | 2.08 (34.94) | 11.11 (12.73) |
  Week 41: number analyzed (Participants) | 6 | 3 | 1 | 4 | 0
  Week 41 | 0.0 (11.79) | 19.44 (12.73) | 16.67 | -2.08 (31.46) |
  Week 49: number analyzed (Participants) | 7 | 3 | 2 | 1 | 0
  Week 49 | 3.57 (13.49) | 16.67 (16.67) | 4.17 (17.68) | 8.33 |

9. Secondary Outcome: Mean Changes From Baseline in the EORTC Brain Cancer Quality of Life Questionnaire (EORTC-QLQ-BN-20)
Description: Health-related quality of life was measured using an EORTC quality of life questionnaire designed specifically for subjects with brain tumors (BN-20). Questionnaires may be completed by the subject or with the assistance of the examiner at baseline prior to initiation of study therapy, and then approximately every 8 weeks while on study treatment (prior to discussing treatment response at each visit, whenever possible). All single questions are answered using a categorical scale (e.g., 1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much) and linearly transformed to 0 to 100 scales with higher scores for a symptom scale representing higher level of symptoms. The evaluation of HRQoL at each timepoint was measured by mean changes from baseline where baseline is the last non-missing value before the administration of MEDI4736 was reported.
Time Frame: Up to 12 months
Population: Number of subjects who completed EORTC Brain Cancer Quality of Life Questionnaire (EORTC-QLQ-BN-20) at baseline and each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
Number analyzed (Participants) | 40 | 31 | 33 | 33 | 22
units on a scale
  Week 9: number analyzed (Participants) | 29 | 14 | 23 | 26 | 10
  Week 9 | 3.63 (8.28) | 5.62 (16.46) | 4.26 (15.95) | 3.50 (15.99) | -2.17 (17.14)
  Week 17: number analyzed (Participants) | 25 | 8 | 14 | 14 | 2
  Week 17 | 0.85 (11.71) | 0.21 (8.93) | -2.55 (18.17) | -4.06 (14.33) | 9.17 (3.54)
  Week 25: number analyzed (Participants) | 20 | 3 | 9 | 5 | 0
  Week 25 | -0.82 (11.12) | -3.33 (8.66) | 3.27 (18.46) | -1.37 (11.80) |
  Week 33: number analyzed (Participants) | 8 | 3 | 4 | 3 | 0
  Week 33 | 6.46 (16.94) | -4.44 (10.05) | -9.39 (16.32) | -17.28 (10.64) |
  Week 41: number analyzed (Participants) | 6 | 2 | 1 | 4 | 0
  Week 41 | 1.94 (18.72) | -5.83 (15.32) | 5.00 | -3.60 (10.38) |
  Week 49: number analyzed (Participants) | 6 | 3 | 2 | 1 | 0
  Week 49 | 5.56 (22.08) | -1.11 (5.36) | 5.83 (5.89) | 2.46 |

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date (i.e., up to 15 months after the first dose of study treatment) are documented, regardless of the causal relationship to study drug. AEs that occur or worsen in severity after the first dose of study treatment are considered treatment emergent (i.e., TEAEs).
Description: AE documentation includes onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms are counted only once per subject at the maximum reported grade.
Arm/Group | Cohort A | Cohort B | Cohort B2 | Cohort B3 | Cohort C
All-Cause Mortality (participants affected / at risk) | 10/40 | 4/31 | 6/33 | 3/33 | 7/22
Serious Adverse Events (participants affected / at risk) | 26/40 | 18/31 | 11/33 | 15/33 | 14/22
Other Adverse Events (participants affected / at risk) | 40/40 | 31/31 | 33/33 | 33/33 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=40) | Cohort B (N=31) | Cohort B2 (N=33) | Cohort B3 (N=33) | Cohort C (N=22)
Headache (Nervous system disorders) | 2 | 2 | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 0 | 1 | 1
Malignant Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4 | 6 | 3 | 6
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 2 | 5 | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Craniotomy (Surgical and medical procedures) | 2 | 3 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 9 | 4 | 2 | 3 | 5
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 0
Brain oedema (Nervous system disorders) | 2 | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 1 | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tumour excision (Surgical and medical procedures) | 4 | 0 | 1 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Biopsy brain (Investigations) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neurologic neglect syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Pyschotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Drowning (General disorders) | 1 | 0 | 0 | 0 | 0
Mass (General disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hallucination, olfactory (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=40) | Cohort B (N=31) | Cohort B2 (N=33) | Cohort B3 (N=33) | Cohort C (N=22)
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 0
Alanine aminotransferase increased (Investigations) | 8 | 4 | 6 | 9 | 4
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 5 | 2
Aphasia (Nervous system disorders) | 11 | 3 | 6 | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 8 | 7 | 2
Aspartate aminotransferase increased (Investigations) | 11 | 4 | 4 | 8 | 1
Asthenia (General disorders) | 2 | 2 | 3 | 0 | 1
Ataxia (Nervous system disorders) | 2 | 3 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 3 | 0
Balance disorder (Nervous system disorders) | 1 | 2 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 2 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2 | 3 | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 6 | 2 | 1 | 1 | 4
Confusional state (Psychiatric disorders) | 6 | 5 | 2 | 2 | 6
Constipation (Gastrointestinal disorders) | 10 | 6 | 4 | 7 | 3
Convulsion (Nervous system disorders) | 5 | 1 | 6 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 6 | 6 | 5
Depression (Psychiatric disorders) | 8 | 2 | 1 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 3 | 6 | 8 | 1
Dizziness (Nervous system disorders) | 10 | 7 | 6 | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 4 | 1 | 0
Dysarthria (Nervous system disorders) | 2 | 2 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 2 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 5 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 5 | 9 | 4 | 3
Fatigue (General disorders) | 29 | 10 | 13 | 18 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1
Gait disturbance (General disorders) | 13 | 10 | 11 | 5 | 5
Headache (Nervous system disorders) | 19 | 12 | 9 | 9 | 8
Hemiparesis (Nervous system disorders) | 4 | 3 | 12 | 3 | 4
Hot flush (Vascular disorders) | 2 | 2 | 1 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 6 | 8 | 5 | 5
Hyperthyroidism (Endocrine disorders) | 4 | 2 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 5 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 5 | 5 | 5
Hypothyroidism (Endocrine disorders) | 3 | 3 | 2 | 3 | 1
Lymphocyte count decreased (Investigations) | 3 | 5 | 0 | 0 | 4
Memory impairment (Nervous system disorders) | 2 | 7 | 2 | 2 | 2
Micturition urgency (Renal and urinary disorders) | 3 | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4 | 2 | 0
Nausea (Gastrointestinal disorders) | 12 | 6 | 5 | 4 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 1 | 0
Oedema peripheral (General disorders) | 4 | 2 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 3 | 4 | 5 | 5 | 2
Platelet count decreased (Investigations) | 2 | 4 | 4 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 2 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 3 | 2 | 1 | 2 | 2
Visual field defect (Nervous system disorders) | 2 | 3 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2 | 1 | 1
Weight decreased (Investigations) | 5 | 2 | 2 | 2 | 1
Agitation (Psychiatric disorders) | 3 | 0 | 2 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 1 | 2 | 0 | 0
Amylase increased (Investigations) | 7 | 1 | 6 | 6 | 0
Anxiety (Psychiatric disorders) | 7 | 0 | 4 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 3 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 3 | 1 | 3 | 1 | 0
Chills (General disorders) | 2 | 0 | 2 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 1 | 5 | 4 | 1
Dry eye (Eye disorders) | 2 | 0 | 2 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 12 | 9 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 2
Facial paresis (Nervous system disorders) | 2 | 0 | 2 | 2 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 3 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Hypertension (Vascular disorders) | 6 | 1 | 8 | 5 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 2 | 1
Insomnia (Psychiatric disorders) | 11 | 1 | 5 | 4 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 2 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 4 | 1
Lipase increased (Investigations) | 11 | 1 | 6 | 5 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 7 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 2 | 4 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 4 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 4 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 5 | 3 | 1
Skin infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 2 | 0
Thyroxine free decreased (Investigations) | 1 | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 5 | 4 | 1
Vision blurred (Eye disorders) | 5 | 1 | 3 | 2 | 1
White blood cell count decreased (Investigations) | 3 | 1 | 2 | 4 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1 | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 1 | 2 | 2
Catheter site pain (General disorders) | 2 | 0 | 0 | 2 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 4
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0 | 2 | 0
Incontinence (Renal and urinary disorders) | 3 | 0 | 0 | 2 | 1
Injection site bruising (General disorders) | 1 | 0 | 1 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0
Tremor (Nervous system disorders) | 6 | 0 | 1 | 2 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 4 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 2 | 0
Irritability (Psychiatric disorders) | 3 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 4 | 2 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 4 | 1 | 1 | 1 | 1
Disturbance in attention (Nervous system disorders) | 3 | 0 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 6 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 3 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 3 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 4 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 3 | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The primary study endpoints have been met; final data will be incorporated upon study completion and availability of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT02336165/Prot_SAP_000.pdf